CLINICAL TRIAL: NCT02049229
Title: Comparison of Titanium-Nitride-Oxide Coated Bio-Active-Stent (Optimax™) to the Drug (Everolimus) -Eluting Stent (Synergy™) in Acute Coronary Syndrome
Acronym: TIDES-ACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital District of Satakunta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA-008
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention; Atherosclerosis
Keywords: Stent; Titanium; drug eluting stent; myocardial infarction; stent thrombosis
MeSH Terms: conditions — Myocardial Infarction; Atherosclerosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OPTIMAX stent (Experimental): Patients randomised to receive titanium-nitride-oxide coated OPTIMAX-stent
  Interventions: Device: percutaneous coronary intervention
- SYNERGY stent (Active Comparator): Patients randomised to receive everolimus-eluting, biabsorabble polymer coated stent
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention — Optimax-stent implantation
  Other Names: Titanium-nitride-oxide coated stent
  Arms: OPTIMAX stent
Device: percutaneous coronary intervention — Synergy stent implantation
  Other Names: Bioabsorbable polymer coated, everolimus-eluting stent
  Arms: SYNERGY stent

SUMMARY:
The purpose of the prospective, randomized and a multicenter trial is to compare clinical outcome in patients presenting with ACS, treated with PCI using Optimax-BAS versus Synergy-EES.

Second objective is to explore whether the Optimax-BAS use is superior compared with Synergy-EES use with respect of hard end points (cardiac death, MI and major bleeding).

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most frequent cause of death, accounting for approximately 13% of all deaths. In western countries, the incidence of ST-segment elevation myocardial infarction (STEMI) is around 77/100 000/year, whereas in patients with non-ST-segment elevation acute coronary syndrome (NSTE-ACS), the incidence is 132/100 000/year. Thus, the incidence of STEMI is decreasing, while there is a concomitant increase in the incidence of NSTE-ACS. NSTE-ACS and STEMI are usually considered to be different entities, but recent reports suggested that the prognosis of either subgroup of MI is similar despite different management strategies. In STEMI, primary percutaneous coronary intervention (PCI) is the recommended reperfusion therapy over fibrinolysis if performed by an experienced team within 2 hours of first medical contact. Treatment of patients with NSTE-ACS is based on their risk of acute thrombotic complications. A clear benefit from early angiography (<48 h) and PCI has been reported in the high-risk patients. However, deferral of interventions does not improve outcome. In addition, routine stenting is recommended on the basis of the predictability of the results and its safety. Consensus has emerged that early PCI use results in favourable outcomes, especially in high-risk patients. The ESC guidelines for NSTE-ACS were updated in 20113 and for STEMI in 2012. Currently, PCI is the preferred reperfusion strategy in patients with both acute STEMI and NSTE-ACS.

Drug-eluting stents (DES) have been shown to reduce in-stent restenosis after PCI compared to bare metal stents (BMS). Over the previous decade, the appearance of first-generation drug-eluting stents (Taxus™, Cypher™) in scene has revolutionized the practice of coronary intervention, resulting in a reduction of restenosis rates by one-half to two-thirds at 5 years follow-up, amounting to roughly 10-15% need for target vessel revascularization following DES at long-term. However, early randomized first-generation-DES trials excluded patients with acute myocardial infarction (MI), even though invasive approach is currently the preferred method for treatment of acute MI. Later randomized trials and meta-analyses of the clinical trials on the use of DES for treatment of acute STEMI demonstrated that the use of DES is safe and improves clinical outcomes mainly by decreasing the risk of re-intervention compared with BMS. However, accumulating evidence from meta-analyses and registries has questioned the long-term safety of first-generation DES, raising concerns about a higher risk of late - and very late - stent thrombosis (ST), a potentially life-threatening complication.

A further step forward was taken with the design of second-generation DES. In SPIRIT I-III trials, everolimus-eluting stent (EES) showed promising mid-term clinical outcome in selected patient groups resulting in FDA approval. Newer, second generation DES are now available in every day practice in interventional cardiology. In this context, Xience-V™-EES significantly reduced late lumen loss, as assessed by angiography, as compared with the paclitaxel-eluting stents (Taxus), with non-inferior rates of a composite outcome of safety and efficacy. Subsequent randomized trials demonstrated that, as compared with first-generation DES, Xience-V-EES was able to reduce both the restenosis and ST rates in overall elective patient population. In Examination trial, Xience-V-EES showed reduced rates of repeat revascularization and ST in STEMI patients when compared with traditional BMS. On the other hand, novel Promus-Element™-EES has showed to be non-inferior when compared with Xience-V-EES in recent all comers-trial. The Promus-Element stent uses the identical drug coating formulation and drug dose density as the Xience-V- stent.

Although, DES delivering antiproliferative drugs from adurable polymer have significantly reduced restenosis compared with BMS, with no apparent increase in the risk of adverse events, durable polymers have been associated with a hypersensitivity reaction, delayed healing, and incomplete endothelialization that may contribute to an increased risk of late (30 days to 1 year) and very late (beyond 1 year) stent thrombosis compared with BMS. A number of stent technologies are being developed in an attempt to modify the proposed mediators of late thrombotic events including bioabsorbable polymers, nonpolymeric stent surfaces, and bioabsorbable stents. Synergy™-EES is a novel Promus-Element stent platform that deliveres everolimus from an ultrathin bioabsorbable polymer applied to the abluminal surface. In the randomized EVOLVE trial, the SYNERGY stent was noninferior to the PROMUS Element stent for the primary angiographic endpoint of in-stent late loss at 6 months. Clinical event rates were low and comparable, with no stent thrombosis observed. These results support the safety and efficacy of the abluminal bioabsorbable polymer SYNERGY EES for the treatment of patients with de novo coronary artery lesions.

The safety of titanium-nitride-oxide-coated bioactive stents (Titan-2™-BAS) has been established in several reports from real-life unselected populations. Interestingly, prospective studies demonstrated an even 'better' outcome with Titan-2-BAS as compared with paclitaxel-eluting stents (Taxus) in high-risk patients with complex coronary lesions, and in patients presenting with acute myocardial infarction (MI). The recent BASE-ACS trial demonstrated that in patients undergoing early PCI for acute coronary syndrome (ACS), the insertion of Titan-2-BAS was non-inferior to Xience-V-EES concerning the occurrence of the primary composite endpoint of MACE at 12 months follow-up. The relative risk ratio of MACE for Titan-2-BAS was 1.07 (a 0.6-percentage-point absolute risk difference) as compared with Xience-V-EES, a difference that met the chief aim of the trial for non-inferiority of Titan-2-BAS in reducing MACE in this patient category. Moreover, albeit not adequately powered to address the individual components of safety and efficacy, non-fatal MI occurred significantly less frequently and ARC-definite ST trended to be lower in the Titan-2-BAS group as compared with the Xience-V-EES group. On the other hand, stent coating with compounds like titanium-nitride-oxide seem to decrease acute surface thrombogenicity, and reduce in-stent restenosis when compared with conventional stainless steel stents. Optimax™ stent is a novel, next generation BAS, in which a thicker layer of titanium-nitride-oxide coating is inserted over the stent struts. The rationale of this is to obtain more efficient and rapid vascular healing at the site of the stent implantation.

After the initial enthusiasm for DES based on their impressive reduction in restenosis, there was increasing concern about an increased risk for late ST. Consequently, the recommendation for the duration of dual antiplatelet therapy with aspirin and clopidogrel (DAPT) was incrementally extended from initially 3 months for Cypher™-DES and 6 months for Taxus™-DES to recently at least 12 months for all DES. Not commonly, cardiologists recommend indefinite DAPT if the patient has no bleeding complications during the first 12 months. The need for long-term DAPT is costly and remains the Achilles' heel of DES; namely increase risk of bleeding complication. Newer generation of stents have shown impressively low ST rates, and therefore the excessive bleeding risk of DAPT is being reconsidered. Current guidelines recommend that oral thienopyridine (clopidogrel, prasugrel or ticagrelol) must be continued for up to 12 months after STEMI, with a strict minimum of 1 month for patient receiving BMS and 6 months for patients receiving DES.

Because early discontinuation of DAPT is recognized as the most potent predictor of DES thrombosis, discussion with the patient regarding the need for and duration of DAPT, and the ability to comply with and tolerate DAPT, is mandatory before DES implantation. When the patient is unable to tolerate or comply with DAPT, as well as when surgery is anticipated within 12 months of DES implantation or when the individual bleeding risk is high, BMS implantation should be preferred. In the attempt to increase biocompatibility of BMS, therefore reducing the risk of ST as well as of restenosis without use of polymer-eluted drugs, various coatings have been used. Among them, diamond-like carbon-coated stent and above-mentioned titanium nitric oxide-coated stent have shown promising results making therefore a point for DAPT duration shorter than the 3 months commonly recommended for BMS.

The purpose of the prospective, randomized and a multicenter trial is to compare clinical outcome in patients presenting with ACS, treated with PCI using Optimax-BAS versus Synergy-EES. Second objective is to explore whether the Optimax-BAS use is superior compared with Synergy-EES use with respect of hard end points (cardiac death, MI and major bleeding).

Long-term (12 months) follow-up of patients presenting with ACS (both STEMI and NSTE-ACS) receiving either Optimax-BAS or Synergy-EES will result in comparable clinical outcome (non-inferiority; MACE including cardiac death, MI and repeat revascularization). Secondly, the strategy of Optimax-BAS use is superior to Synergy-EES use during the 18 months of follow-up in hard end points (superiority; cardiac death, MI and major bleeding).

ELIGIBILITY:
Inclusion Criteria:

A) Patients presenting with non ST-elevation acute coronary syndrome:

Ischemic symptoms suspected to represent a non-ST-elevation acute coronary syndrome (UAP / NSTE-MI) defined as:

New onset of characteristic ischemic chest pain occurring at rest or within minimal exercise (lasting longer than 10 minutes) and planned to be managed with an invasive strategy, AND at least one of the following;

* ECG changes compatible with new ischemia (ST depression of at least 1mm or transient ST elevation or ST elevation of ≤ 1mm or T wave inversion greater than 2 mm in at least 2 contiguous leads).
* Already elevated troponin I or T above the upper limit of normal.
* Patients > 60 years of age with normal ECG at admission are eligible provided there is a high degree of certainty that patient's presenting symptoms are due to myocardial ischemia. These patients must have documented evidence of previous coronary artery disease (CAD) with at least one of the following:

Previous MI Previous PCI or CABG Positive exercise test Other evidence of CAD

B) Patients presenting with ST-elevation myocardial infarction (STEMI)

Ischemic symptoms suspected to represent ST-elevation myocardial infarction defined as:

Patients presenting with sign or symptoms of acute MI and planned to be managed with an invasive strategy with intent to perform a PCI during the index hospitalization.

ECG changes compatible with STEMI: persistent ST-elevation (>2mm in two contiguous leads or > 1mm in at least two limb leads), or new left bundle branch block, or Q-wave in two contiguous leads.

II) Written informed consent

Exclusion Criteria:

* Age < 18 years
* Expected survival < 1 year
* Allergy to aspirin, clopidogrel, prasugrel or ticagrelol
* Allergy to heparins, glycoprotein IIb/IIIa inhibitors or bivalirudin
* Allergy to everolimus
* Active bleeding or significant increased risk of bleeding
* Stent length longer than 28 mm needed
* Stent diameter > 4.0 mm needed
* Previous coronary artery bypass surgery (CABG)
* Aorto-ostial lesion
* Previous coronary stenting of the target vessel
* Thrombolysis therapy
* Cardiogenic shock
* Planned surgery within 12 months of PCI unless the dual antiplatelet therapy could be maintained throughout the perisurgical period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 months
  The primary end point (MACE) is the composite of cardiac death, myocardial infarction (MI) and target lesion revascularization (TLR) during 12 months of follow-up (non-inferiority).
cardiac death, any myocardial infarction and major bleeding | 18 months
  Co-Primary end point is the composite of during 18 months of follow-up (superiority).

SECONDARY OUTCOMES:
Composite of cardiac death, MI, stent thrombosis and TLR | 1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years.
  Composite of cardiac death, MI, stent thrombosis and TLR
Cardiac death or myocardial infarction | Cardiac death or myocardial infarction
  1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years.
Stent thrombosis | Stent thrombosis
  1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years
All cause death | All cause death
  1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years.
TLR | Target lesion revascularization
  1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years.
TVR | Target vessel revascularization
  1, 6, 12 and 18 months, and at 2, 3, 4 and 5 years.
Major Bleeding (ARC-definition) | Major Bleeding (ARC-definition)
  1, 6, 12 and 18 months.

CONTACTS AND LOCATIONS:
Locations (6):
- Finland (6):
  - Heart Center, Helsinki University Hospital, Helsinki
  - Kokkola Central Hospital, Kokkola
  - Heart Center, Kuopio University Hospital, Kuopio
  - Dep.Of Cardiology, Oulu University Hospital, Oulu
  - Heart Center, Satakunta Central Hospital, Pori
  - Heart Center, Turku University Hospital, Turku

REFERENCES:
- [Derived] Bouisset F, Sia J, Mizukami T, Karjalainen PP, Tonino PAL, Pijls NHJ, Van der Heyden J, Romppanen H, Kervinen K, Airaksinen JKE, Lalmand J, Frambach P, Roza da Costa B, Collet C, De Bruyne B; TIDES-ACS Study Group. Titanium-Nitride-Oxide-Coated vs Everolimus-Eluting Stents in Acute Coronary Syndrome: 5-Year Clinical Outcomes of the TIDES-ACS Randomized Clinical Trial. JAMA Cardiol. 2023 Jul 1;8(7):703-708. doi: 10.1001/jamacardio.2023.1373. PMID 37203243
- [Derived] Tonino PAL, Pijls NHJ, Collet C, Nammas W, Van der Heyden J, Romppanen H, Kervinen K, Airaksinen JKE, Sia J, Lalmand J, Frambach P, Penaranda AS, De Bruyne B, Karjalainen PP; TIDES-ACS Study Group. Titanium-Nitride-Oxide-Coated Versus Everolimus-Eluting Stents in Acute Coronary Syndrome: The Randomized TIDES-ACS Trial. JACC Cardiovasc Interv. 2020 Jul 27;13(14):1697-1705. doi: 10.1016/j.jcin.2020.04.021. PMID 32703593
- [Derived] Colkesen EB, Eefting FD, Rensing BJ, Suttorp MJ, Ten Berg JM, Karjalainen PP, Van Der Heyden JA. TIDES-ACS Trial: comparison of titanium-nitride-oxide coated bio-active-stent to the drug (everolimus)-eluting stent in acute coronary syndrome. Study design and objectives. Minerva Cardioangiol. 2015 Feb;63(1):21-9. PMID 25670057